CLINICAL TRIAL: NCT02485990
Title: An Open Label Dose Escalation/Expansion Study of Tremelimumab Alone or Combined With Olaparib for Recurrent or Persistent EOC (Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma)
Brief Title: Study of Tremelimumab Alone or Combined With Olaparib for Patients With Persistent EOC (Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawal of sponsor support
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: AstraZeneca (Industry); MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J15113; IRB00064379 (Other: JHM IRB)
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Primary Peritoneal Carcinoma
Keywords: Fallopian Tube; Epithelial Ovarian; EOC
MeSH Terms: interventions — tremelimumab; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: Tremelimumab Alone (Experimental): 25 patients will receive tremelimumab alone at 10 mg/kg IV every 4 weeks for 7 doses then every 12 weeks until disease progression.
  Interventions: Drug: Tremelimumab
- Arm B1: DESE Tremelimumab and Olaparib (Experimental): 18 patients will receive tremelimumab (3 or 10 mg/kg IV) every 4 weeks for 7 doses then every 12 weeks and olaparib (150 or 300 mg orally twice a day) until disease progression.
  Interventions: Drug: Tremelimumab; Drug: Olaparib
- Arm B2: Tremelimumab and Olaparib (Experimental): 25 patients will receive tremelimumab (every 4 weeks for 7 doses then every 12 weeks) and olaparib (daily) until disease progression. Dose of tremelimumab and olaparib will be determined during the DESE (Arm B1).
  Interventions: Drug: Tremelimumab; Drug: Olaparib

INTERVENTIONS:
Drug: Tremelimumab
Drug: Olaparib
  Other Names: LYNPARZA
  Arms: Arm B1: DESE Tremelimumab and Olaparib; Arm B2: Tremelimumab and Olaparib

SUMMARY:
This study will be looking at what dose of tremelimumab and olaparib is safe and effective in patients with persistent EOC (Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma).

DETAILED DESCRIPTION:
This clinical trial was initially intended to be a Phase 1/2 trial, but the trial never moved forward to Phase 2 prior to termination.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Age ≥ 18 years
3. Recurrent or persistent EOC (epithelial ovarian, fallopian tube or primary peritoneal carcinoma)
4. Have archival tissue or willingness to undergo a tumor biopsy
5. Have measurable disease
6. Have had one prior taxane-platinum-based chemotherapeutic regimen
7. Have had a treatment-free interval following platinum-based therapy of less than 12 months, have progressed during platinum-based therapy, or had persistent disease after a platinum-based regimen
8. Have received hormonal therapy
9. ECOG Performance Status of 0 to 1
10. Ability to take oral medications
11. HIV, HTLV-1, HBV, and HCV negative
12. Adequate organ and bone marrow function as defined by study-specified laboratory tests
13. Normal blood coagulation parameters
14. Life expectancy greater than 16 weeks
15. Must use acceptable form of birth control through the study and for 28 days after final dose of study drug
16. Willing and able to comply with study procedures

Exclusion Criteria:

1. Prior therapy with an anti-CTLA-4 antibody or PARP inhibitor
2. Active infection requiring antibiotics
3. Active autoimmune disease
4. Active and uncontrolled intercurrent illness
5. History of other cancers within the past 5 years
6. Systemically active steroid use
7. Receiving systemic chemotherapy or radiotherapy within 4 weeks prior to the first dose of study drug
8. Use of ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir
9. Requirement for chronic parenteral hydration/nutrition
10. Vaccination with live attenuated vaccine within 1 month prior to first dose of study drug
11. Patients with untreated brain metastases, treated brain metastases that are not stable, leptomeningeal disease, or seizures uncontrolled with standard medical therapy
12. Patients with myelodysplastic syndrome/acute myeloid leukaemia
13. History of diverticulitis
14. History of bleeding disorder or diathesis.
15. Serious or nonhealing wound, ulcer, bone fracture, or osteonecrosis of the jaw
16. Major surgical procedure within 28 days of study enrollment, or anticipated while on study.
17. Pregnant or breast feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Adverse events as a measure of the safety and tolerability profile of tremelimumab in combination with olaparib | 4 years
  Number of participants experiencing study drug-related dose limiting toxicities (DLTs). Dose escalation (phase I) portion of the trial only.
Fold change from baseline in the ratio of peripheral CD4+ICOShi T cells and Regulatory T cells | 4 years
  Dose escalation (phase I) portion of the trial only.
Maximum Tolerated Dose (MTD) of tremelimumab combined with olaparib | 4 years
  Dose escalation (phase I) portion of the trial only.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) Rate at 6 months by RECIST | 6 months
  PFS rate is defined as the percentage of patients with disease progression (PD or relapse from CR as assessed using RECIST 1.1 criteria) or death due to any cause at 6 months. Per RECIST 1.1 criteria, Complete Response (CR) = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Progression Free Survival (PFS) Rate at 6 months by irRECIST | 6 months
  PFS rate is defined as the percentage of patients with disease progression (irPD or relapse from irCR as assessed using irRECIST criteria) or death due to any cause at 6 months. Per irRECIST criteria, irCR = disappearance of all lesions, irPR is =>30% decrease in tumor burden, irPD is >20% increase in tumor burden compared with nadir, irSD is <30% decrease in tumor burden compared with baseline cannot be established nor <20% increase compared with nadir. Estimation based on the Kaplan-Meier curve.
Objective Response Rate (ORR) by RECIST | 4 years
  Objective Response Rate (ORR) is defined as the percentage of patients achieving a complete response (CR) or partial response (PR) based on RECIST 1.1 criteria. Per RECIST 1.1 criteria, CR = disappearance of all target lesions and PR is =>30% decrease in sum of diameters of target lesions.
Objective Response Rate (ORR) by irRECIST | 4 years
  Objective Response Rate (irORR) is defined as the percentage of patients achieving a complete response (irCR) or partial response (irPR) based on irRECIST criteria. Per irRECIST criteria, irCR = disappearance of all lesions and irPR is =>30% decrease in tumor burden.
Duration of Response by RECIST | 4 years
  Number of months from the start date of PR or CR (whichever response is recorded first) and subsequently confirmed to the first date that recurrent or progressive disease or death is documented. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, and PD is >20% increase in sum of diameters of target lesions.
Duration of Response by irRECIST | 4 years
  Number of months from the start date of irPR or irCR (whichever response is recorded first) and subsequently confirmed to the first date that recurrent or progressive disease or death is documented. Per irRECIST criteria, irCR = disappearance of all lesions, irPR is =>30% decrease in tumor burden, and irPD is is >20% increase in tumor burden compared with nadir.
Disease Control Rate (DCR) | 4 years
  DCR is defined as the number of patients achieving a complete response (CR) or partial response (PR) or stable disease (SD) based on RECIST 1.1 criteria at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, PD is >20% increase in sum of diameters of target lesions, SD is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Progression-Free Survival (PFS) | 4 years
  PFS is defined as the number of patients with disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Overall Survival (OS) | 4 years
  OS will be measured from date of first dose until death or end of followup (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Gaillard, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States